CLINICAL TRIAL: NCT05929313
Title: A Prospective, Multicenter, Randomized Controlled, Non- Inferiority Trial to Evaluate the Effectiveness and Safety of the Scoreflex TRIO High-pressure Tri-wire Scoring Balloon Catheter for Balloon Dilatation of Coronary Artery Stenosis
Brief Title: Scoreflex TRIO - Scoring PTCA Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OrbusNeich (Industry)
Collaborators: CCRC Medtech (Shanghai) Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SFT-2022-001
Record Dates: First submitted 2023-06-23; First posted 2023-07-03 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Coronary Arteriosclerosis
Keywords: Coronary Artery Disease; Coronary Disease; Myocardial Ischemia; Heart Diseases; Arteriosclerosis; Cardiovascular Diseases
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease; Myocardial Ischemia; Heart Diseases; Arteriosclerosis; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OrbusNeich Scoreflex TRIO (Experimental): OrbusNeich Scoreflex TRIO Scoring PTCA catheters
  Interventions: Device: OrbusNeich Scoreflex TRIO
- OrbusNeich Scoreflex NC (Active Comparator): OrbusNeich Scoreflex NC Scoring PTCA catheters
  Interventions: Device: OrbusNeich Scoreflex NC

INTERVENTIONS:
Device: OrbusNeich Scoreflex TRIO — To dilate coronary arteries during the subject's index procedure with Scoreflex TRIO Scoring PTCA catheters
  Arms: OrbusNeich Scoreflex TRIO
Device: OrbusNeich Scoreflex NC — To dilate coronary arteries during the subject's index procedure with Scoreflex NC Scoring PTCA catheters
  Arms: OrbusNeich Scoreflex NC

SUMMARY:
To evaluate the acute safety and device procedural success of the Scoreflex TRIO Scoring PTCA catheters versus Scoreflex NC Scoring PTCA catheters in subjects with stenotic coronary arteries during percutaneous coronary intervention.

DETAILED DESCRIPTION:
This is a prospective, multi-center, open-label, non-inferiority, randomized controlled trial which plans to enroll 210 subjects. All subjects enrolled will be randomly assigned to the test group (n=105) and the control group (n=105). Subjects in the test group and the control group will receive Scoreflex TRIO Scoring PTCA catheters and Scoreflex NC Scoring PTCA catheters respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and≤ 80.
2. Volunteer to participate in this trial and provide the written informed consent.
3. Subjects must have a single or double vessel coronary artery disease (CAD) and clinical evidence of ischemic heart disease, such as CAD, stable / unstable angina or silent ischemia, need percutaneous coronary intervention.

   Angiographic Inclusion Criteria
4. Subject must have de novo or restenotic lesion(s) in native coronary arteries, including in-stent restenosis suitable for percutaneous coronary intervention.
5. A maximum of two lesions that needed to be treated and they are located in two coronary arteries, including at least one target lesion, in up to two coronary arteries.
6. Target lesion must have a reference vessel diameter (RVD) between 1.75 and 4.0 mm by visual estimation.
7. Target lesion(s) must have a diameter stenosis of ≥70% by visual estimation.
8. The non-target lesion must be located in different coronary artery from the Target lesion. Treatment of non-target lesion, if any, must be completed prior to treatment of target lesion and must be deemed a clinical angiographic success as visually assessed by the physician.

Exclusion Criteria:

1. STEMI or NSTEMI within 7 days of study screening.
2. A serum creatinine level > 2.0 mg/dl within 7 days prior to index procedure.
3. Cerebrovascular accident (CVA) within the past 6 months.
4. Active peptic ulcer or active gastrointestinal (GI) bleeding within the past 6 months.
5. Left ventricular ejection fraction (LVEF) <30% (LVEF may be obtained at the time of the index procedure if the value is unknown, if necessary)
6. Subject with a known hypersensitivity or contraindication to aspirin, heparin, bivalirudin, anti-platelet medications,
7. Subject is known to be allergic to the ingredients of the test product and the sensitivity to contrast media.
8. Subject with known pregnancy or is nursing. Women of child-bearing potential should have a documented negative pregnancy test within 7 days before index procedure.
9. Planned or actual target lesion treatment with an unapproved device, atherectomy, laser, cutting balloon or thrombectomy during the index procedure.
10. Subjects who are participating in clinical research of other drugs and devices.
11. Other conditions assessed by the investigator as inappropriate to participate in this trial.

    Angiographic Exclusion Criteria
12. Target lesion longer than 30 mm by visual estimation.
13. Extreme angulation (90º or greater) proximal to or within the target lesion.
14. Target lesion located within an arterial or saphenous vein graft or graft anastomosis
15. Previous percutaneous intervention of lesions in a target vessel (including side branches) conducted within 9 months before the study procedure and located within 10 mm from the current target lesion.
16. Target lesion demonstrating severe dissection prior to planned deployment of the investigational device.
17. Unprotected left main coronary artery disease.
18. Coronary artery spasm of the target vessel in the absence of a significant stenosis.
19. Target lesion with angiographic presence of probable or definite thrombus.
20. Target lesion involves a bifurcation requiring treatment with more than one stent or pre-dilatation of a side branch >2.0 mm in diameter.
21. Non-target lesion to be treated during the index procedure meets any of the following criteria:

    * Located within a bypass graft (venous or arterial)
    * Left main location
    * Chronic total occlusion
    * Involves a bifurcation (e.g., bifurcations requiring treatment with more than 1 stent)
    * Treatment not deemed a clinical angiographic success

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2023-04-27 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-29 (Actual)

PRIMARY OUTCOMES:
Rate of device Procedural Success | Peri-procedural (at Day 0)
  Device procedural success consisting of the following:
  * Successful delivery, inflation, deflation, and withdrawal of the device
  * No evidence of vessel perforation, flow limiting dissection (grade C or higher) or reduction in Thrombolysis In Myocardial Infarction (TIMI) flow from baseline as related to the devices
  * Residual stenosis of target lesion <50% after balloon angioplasty, Final TIMI flow grade of 3 at the conclusion of the percutaneous coronary intervention (PCI) procedure

SECONDARY OUTCOMES:
Improvement in Minimum Lumen Diameter (MLD) following use of Scoreflex NC catheter (measured by QCA). | Peri-procedural (at Day 0)
  Improvement in MLD is defined as MLD post use of Scoreflex as greater than MLD from baseline.
In-hospital Major Adverse Cardiac Events (MACE) | Endpoints will be measured through hospital discharge (expected to be within 24 hours)
  In-hospital Major Adverse Cardiac Events (MACE), a composite of: Cardiac death, Myocardial Infarction (MI), Target Lesion Revascularization (TLR), clinically driven.
Device-oriented target lesion failure (TLF) | 30 days
  The device-oriented target lesion failure (TLF) is defined as a composite of cardiac death, target vessel myocardial infarction (MI), and ischemia-driven target lesion revascularization (i-TLR)
Patient-oriented composite endpoint | 30 days
  The patient-oriented composite endpoint includes all-cause death, all MIs, or any revascularization.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Bo Ge, MD, Principal Investigator — Fudan University
Locations (4):
- China (4):
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Tong Ren Hospital Shanghai Jiao Tong University School of Medicine, Shanghai
  - Zhongshan Hospital Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: No